CLINICAL TRIAL: NCT03260972
Title: An Evaluation of Intraabdominal Chloroprocaine During Cesarean Delivery and Its Effect on Postoperative Pain and Nausea; a Randomized Controlled Trial & Pharmacokinetic-pharmacodynamics (PKPD) Analysis.
Brief Title: Intraabdominal Chloroprocaine During Cesarean Delivery for Pain Control
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn by IRB
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00129099
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cesarean Section Complications; Pain
MeSH Terms: conditions — Pain | interventions — chloroprocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients admitted for cesarean section and meeting inclusion criteria will be approached for consent. Consented patients will then be randomized into two groups.
  Group 1: (intraabdominal chloroprocaine administration): These participants will have intraabdominal chloroprocaine administration at the time of cesarean section before fascial closure.
  Group 2: (Intraabdominal instillation of placebo (sterile water): These participants will have placebo (normal saline) administered at the time of cesarean section before fascial closure. Cesarean section will proceed traditionally, including fascial and skin closure.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator and patients will be masked from the treatment options. The care providers will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chloroprocaine arm (Active Comparator): 20 mls of Chloroprocaine Hcl 2% Inj (1 vial containing 400mg/20 mls of chloroprocaine) will be instilled into the abdomen prior to fascia closure.
  Interventions: Drug: Chloroprocaine Hcl 2% Inj
- Normal saline arm (Placebo Comparator): 20 mls of normal saline will be instilled into the abdomen prior to fascia closure.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Chloroprocaine Hcl 2% Inj — 20 mls of Chloroprocaine Hcl 2% Inj (1 vial containing 400mg/20 mls of chloroprocaine) will be instilled into the abdomen prior to fascia closure.
  Other Names: Nesacaine
  Arms: Chloroprocaine arm
Drug: Normal saline — 20 mls of normal saline will be instilled into the abdomen prior to fascia closure.
  Arms: Normal saline arm

SUMMARY:
Objective The objective of this study is to test the hypothesis that instillation of intra-abdominal chloroprocaine during cesarean deliveries is associated with decreased postoperative pain and nausea compared to placebo, without increasing intraoperative and postoperative complications.

Methods The investigators plan to randomize about 150 women undergoing primary and repeat cesarean deliveries to intra-abdominal chloroprocaine versus placebo prior to abdominal closure. Women will be excluded if they have ascertained or presumptive hypersensitivity to the ester type and major anesthetics; if they have chronic pelvic pain or if they refuse to participate in the study. The investigators' primary outcome measure will be postoperative pain as measured by visual analogue scale (VAS) at 1 hour after skin closure. Secondary outcomes will include objective pain as measured by VAS at 2, 6, 24 and 48 hours at rest and during mobilization, adverse effects of chloroprocaine (gastrointestinal side effects, pruritus), concomitant analgesic requirement, hospital readmissions and length of hospital stay. Analysis will follow the intention-to-treat principle.

The investigators will also be studying the concentration/effect (PKPD) relationship of chloroprocaine use for pain control in the postpartum period. The time courses of the plasma concentrations of chloroprocaine will be analyzed with mixed effects pharmacokinetic-pharmacodynamic (PKPD).

DETAILED DESCRIPTION:
Postoperative pain relief is an important consideration during and after cesarean section. Although many different methods have been described for proper pain relief, it remains not sufficient and satisfactory in some patients.1,2 The overprescribing of opioids has reached a critical level worldwide, and cesarean section may be the trigger for long-term opioid use in many patients.1,2,3 The optimal strategy for perioperative pain control consists of multimodal therapy to minimize the need for opioids, with the goals of perioperative pain management being to relieve suffering, achieve early mobilization after surgery, reduce length of hospital stay, and achieve patient satisfaction. Currently, most obstetricians use a combination of opioids and NSAIDs for pain control postpartum. These pain control regimens take into account medical, psychological, and physical condition of women, age, level of fear or anxiety, allergies and personal preference at the time of cesarean section. Due to several aspects such as maternal and neonatal wellbeing, postoperative pain relief in cesarean delivery is crucial. Therefore, providing a proper regimen with very quick onset of action, devoid of renal or gastrointestinal complications, and devoid of complications of neonatal abstinence syndrome (NAS) becomes necessary.

Local anesthetics have been extensively used at the time of cesarean section. Chloroprocaine (Nesacaine) is an ester-type local anesthetic (active ingredient - benzoic acid, 4-amino-2-chloro-2-(diethylamino) ethyl ester, monohydrochloride that has been used as an anesthetic and analgesic in obstetrics & gynecology. It has a rapid onset time of action (usually within 6 to 12 minutes; 9.6 min ± 7.3 min at 40 mg dose; 7.9 min ± 6.0 min at 50 mg dose) and a motor block action lasting for 40 minutes to 2 hours.4 Chloroprocaine, like other local anesthetics, blocks the generation and the conduction of nerve impulses, presumably by increasing the threshold for electrical excitation in the nerve, by slowing the propagation of the nerve impulse and by reducing the rate of rise of the action potential. In general, the progression of anesthesia is related to the diameter, myelination and conduction velocity of affected nerve fibers.

The rate of intra-abdominal chloroprocaine absorption is dependent upon the total dose and concentration administered and the presence or absence of epinephrine in the anesthetic injection. Epinephrine usually reduces the rate of absorption and plasma concentration of local anesthetics and is sometimes added to local anesthetic injections in order to prolong the duration of action. Various pharmacokinetic parameters of chloroprocaine can be significantly altered by the presence of hepatic or renal disease, addition of epinephrine, factors affecting urinary pH, renal blood flow, and the age of the patient. Chloroprocaine is rapidly metabolized in plasma by hydrolysis of the ester linkage by pseudocholinesterase. The hydrolysis of chloroprocaine results in the production of ß-diethylaminoethanol and 2-chloro-4-aminobenzoic acid, which inhibits the action of the sulfonamides. The kidney is the main excretory organ for chloroprocaine and its metabolites. Urinary excretion is affected by urinary perfusion and factors affecting urinary pH. Due to its short duration of action, favorable safety profile, and very low toxicity, it has been used extensively for spinal anesthesia at the time of cesarean section.5,6 It has also been used for skin infiltration to reduce pain post cesarean section in patients who cannot receive spinal analgesia due to contraindications.7 However, despite its advantages as an analgesic and anesthetic, it has never clinically evaluated to be used intra-abdominally at the time of cesarean section. Although its occasional use has been considered and employed in certain clinical circumstances, clinical evaluation has not been attempted.

The goal of this study is to employ a well-designed randomized controlled clinical trial to compare the efficacy of intraabdominal chloroprocaine administration versus placebo (sterile saline) for pain control at the time of cesarean section. The investigators hypothesize that intra-abdominal chloroprocaine administration at the time of cesarean delivery is associated with decreased postoperative pain and nausea compared to non-administration of chloroprocaine. Patients admitted for cesarean section and meeting inclusion criteria will be approached for consent. Consented patients will then be randomized into two groups.

Group 1: (intraabdominal chloroprocaine administration): These participants will have intraabdominal chloroprocaine administration at the time of cesarean section before fascial closure.

Group 2: (Intraabdominal instillation of placebo (sterile saline): These participants will have placebo (sterile saline) administered at the time of cesarean delivery before fascial closure. Cesarean delivery will continue traditionally, including fascial and skin closure.

Assignment will be performed by opening a sequentially numbered opaque envelope containing computer-randomized individual allocations. The envelope will be opened by the circulation nurse in the operating room and silently viewed by the surgeons prior to surgery. Instructions will be given to not verbalize the treatment arm revealed. The original randomization will be performed by research staff before the initiation of the study using a random number table generator, and the participants will be blinded to treatment once assigned. Information regarding basic demographic data, interventions during the cesarean delivery and postpartum course will be obtained from the participant's charts after discharge from the hospital. The patients will be assessed for pain control, nausea and vomiting after cesarean section. The protocol for labor management and fetal monitoring will be the same for both groups, including continuous electronic fetal monitoring prior to delivery.

Both groups will undergo inspection of the uterine incision, with or without closure of the vesicouterine peritoneum (bladder flap), abdominal peritoneum, or rectus muscles per attending preference. Both groups will undergo standard closure of the abdominal fascia, consisting of suturing with a running non locking delayed absorbable suture. Irrigation of the subcutaneous tissues superior to the closed fascia will be performed in both groups. Staples or absorbable suture will be used for skin closure. In addition, all participants will receive a standardized dose of 1-2 g cefazolin intravenously as antibiotic prophylaxis before the start of surgery. Participants with cefazolin allergy will receive 900 mg clindamycin.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a singleton or multiple pregnancies, vertex or breech presentation presenting to our labor and delivery unit for an elective cesarean section will be eligible for participation.

Exclusion Criteria:

* Women will be excluded if any of the following criteria are encountered: Allergy against local anesthetics - ascertained or presumptive hypersensitivity to the ester type and major anesthetics; chronic pelvic pain and refusal to participate in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) at 1 hour after skin closure | Immediately following cesarean section to 1 hour after skin closure
  Our primary outcome measure will be postoperative pain as measured by visual analogue scale (VAS) at 1 hours after skin closure (sitting in an upright position and movement of lower extremities) after cesarean section. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient selects a whole number (0-10 integers) that best reflects the intensity of their pain, with 0 being the best pain and 10 being the worst pain.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) at 2, 6, 24 and 48 hours at rest and during mobilization | 2, 6, 24 and 48 hours after cesarean section
  Visual analogue scale (VAS) at 2, 6, 24 and 48 hours at rest and during mobilization. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient selects a whole number (0-10 integers) that best reflects the intensity of their pain, with 0 being the best pain and 10 being the worst pain.
Adverse effects of chloroprocaine (gastrointestinal side effects, pruritus) | Day 0 to 2 weeks after delivery
  An adverse effect is an undesired harmful effect resulting from chloroprocaine use. Adverse effects of chloroprocaine include gastrointestinal (nausea, vomiting), dizziness, rash, itching, redness and anxiety.
Concomitant analgesic requirement | Day 0 to 4 weeks after delivery
  The patients will be evaluated for increased analgesic requirement after use of chloroprocaine or placebo. The total amount of analgesia used will be recorded.
Hospital readmissions for pain | Day 0 to 6 weeks after delivery
  A hospital readmission for pain is an episode when a patient who had been adequately pain controlled is discharged from a hospital is admitted again within a specified time interval for poor pain control.
Length of hospital stay | Day 0 to 1 week after delivery
  This is defined as the number of days the patient stays in the hospital after cesarean section.

CONTACTS AND LOCATIONS:
Overall Officials: Ahizechukwu Eke, MD MPH, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No
No personal patient data will be shared with other researchers. The final de-identified manuscript will be published.